CLINICAL TRIAL: NCT00201617
Title: Short-term and Long-term Efficacy of the BAHA for Single Sided Deafness
Brief Title: Efficacy of the Bone-anchored Hearing Aid for Unilateral Deafness
Status: Completed | Type: Observational
Sponsor: The New York Eye & Ear Infirmary (Other)
Collaborators: The Jacob and Valeria Langeloth Foundation (Other)
Other Study IDs: 03.33; 000303
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Unilateral Deafness
Keywords: Unilateral hearing loss; Unilateral deafness; Bone anchored hearing aid
MeSH Terms: conditions — Hearing Loss, Unilateral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: normal hearing sensitivity
- 2: Unilateral deafness who are implanted with a Bone Anchored Hearing Aid
  Interventions: Device: Bone-anchored hearing aid

INTERVENTIONS:
Device: Bone-anchored hearing aid
  Groups: 2

SUMMARY:
The purpose of this 3-year prospective investigation is to examine the short-term and long-term (1 year)efficacy of the bone-anchored hearing aid (BAHA) in adults with single sided deafness

DETAILED DESCRIPTION:
Limited studies have been done on the BAHA in adults with single sided (sensorineural) deafness, and these studies have evaluated only short-term efficacy at one month post implantation. The findings of the limited number of studies to date on the BAHA with single sided deafness demonstrate that the BAHA improves understanding in noisy or group situations and understanding conversation when addressed by a speaker on the side of the bad ear and most users have judged the BAHA to have at least satisfactory benefit. But conflicting findings have been obtained regarding whether the BAHA improves the ability to locate the source of a sound. Additionally, no studies have been done to see whether the magnitudes of the improvements seen at one month post implantation increase over time because of learning effects or brain plasticity.

This investigation will show whether the previously reported BAHA benefits at one month post BAHA sound processor fitting, related to speech recognition in noise and subjective satisfaction, persist at one year, and whether learning effects increase the magnitudes of these benefits from one month to one year post BAHA sound processor fitting. This long-term investigation also attempts to resolve the conflicting findings pertaining to the BAHA effect on localization abilities.

Subjects with hearing impairment will comprise 20 adults with single sided deafness who consent to remediation with the BAHA.In order to see how the adults with unilateral hearing loss will differ from the normal-hearing subjects over time, a control group of 20 normal-hearing individuals also will be evaluated over time, to see how closely the results of the unilateral deafness group approximate the results of the normal individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Adult-onset deafness
2. Deafness is unilateral - complete or near complete

Exclusion Criteria:

1. the presence of a developmental disorder or mental retardation;
2. history of drug abuse;
3. psychiatric disease;
4. inability to follow instructions or to participate in follow-up appointments
5. inability to use the BAHA
6. lack of osseo-integration -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
HINT score | Pre-BAHA, 3 mos post BAHA, 6 mos post BAHA, and 1 year post BAHA
  Hearing in Noise Test
CNC score | Pre-BAHA, 3 mos post BAHA, 6 mos post BAHA, and 1 year post BAHA
  Consonant-nucleus-consonant speech-recognition test
Localization | Pre-BAHA, 3 mos post BAHA, 6 mos post BAHA
  Localization in sound field test

SECONDARY OUTCOMES:
Abbreviated Profiles of Hearing Aid Benefit | 3 months post BAHA, 6 months post BAHA, 1 year post BAHA
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Linstrom, MD, Principal Investigator — New York Eye & Ear Infirmary; Carol A Silverman, PhD, MPH, Principal Investigator — New York Eye & Ear Infirmary
Locations (1):
- New York Eye & Ear Infirmary, New York, New York, United States